CLINICAL TRIAL: NCT00836121
Title: Case Report of a 39 Years Old Man That Has Been Cured by a Total Resection of a Anterior Mediastinum Teratoma.
Brief Title: Anterior Mediastinum Teratoma: A Case Report
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina de Catanduva (Other)
Responsible Party: Stella Mariana Ferreira Giolo, Faculdade de Medicina de Catanduva
Other Study IDs: FAMECA2009; SMFG2009
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Teratoma
Keywords: Teratoma; Mediastinum
MeSH Terms: conditions — Teratoma

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- tumor
  Interventions: Procedure: right thoracotomy

INTERVENTIONS:
Procedure: right thoracotomy — complete surgical resection

SUMMARY:
The investigators report a case of a 39-year-old man who presented an anterior mediastinal cystic mature teratoma. Those kind of tumor contain elements derived from more than one of the three primary germ layers (ectoderm, mesoderm, endoderm), frequently arranged in a haphazard manner. They arise from totipotent cells and, therefore, are primarily found in gonads, and more rarely in primitive cells kidnapped in other parts of the body. The tissues are immature to well differentiated and foreign to the anatomic site. Mature teratomas are either cystic or solid, although the cystic presentation predominates in gonadal sites. Benign teratomas are the most common mediastinal germ cell tumor, accounting 70% of the mediastinal germ cell tumors in children and 60% of those in adults. Immature teratomas are potentially malignant tumors; their prognosis is influenced by the anatomic site of the tumor, patient age, and the fraction of the tumor that is immature. Treatment of benign mediastinal teratoma includes complete surgical resection, with results in a excellent long-term cure rates. Complete resection of teratomas should be the goal of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mediastinum teratoma

Exclusion Criteria:

* Tumor absent

Ages: 39 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
cure | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stella MF Giolo, student, Principal Investigator — Faculdade de Medicina de Catanduva
Locations (1):
- Faculdade de medicina de Catanduva, Catanduva, São Paulo, Brazil